CLINICAL TRIAL: NCT05389657
Title: Dissemination and Implementation of Family-Based Treatment in Publicly-Funded Clinics: Optimizing Provider Training in Eating Disorders (OPTED)
Brief Title: Optimizing Provider Training in Eating Disorders (OPTED)
Acronym: OPTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5K23MH120347 (NIH); 5K23MH120347 (NIH)
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
Keywords: Training; Eating disorders; Family based treatment; Medicaid; Community mental health; Children and adolescents; Mental health clinicians
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based training (Experimental): Web-based training will provide online training primarily focused on family-based treatment and appropriate adaptations to the treatment model.
  Interventions: Behavioral: Web-based training
- Live training (Active Comparator): Live training will include two days of expert-led live training (via zoom). The content of the training will be similar to that provided in web-based training, primarily focused on family-based treatment and appropriate adaptations to the treatment model.
  Interventions: Behavioral: Live training

INTERVENTIONS:
Behavioral: Web-based training — Web-based training will be divided into training modules that will be completed by participants over the course of 6-8 weeks. Training will include didactic training videos, knowledge checks, example sessions, and a library of resources.
  Arms: Web-based training
Behavioral: Live training — The live training will be delivered by two trainers over the course of two days via Zoom.
  Arms: Live training

SUMMARY:
This is a randomized controlled trial for mental health clinicians comparing two methods of training in family-based treatment (FBT) for restrictive eating disorders.

DETAILED DESCRIPTION:
This is a randomized controlled trial for mental health clinicians comparing two methods of training in family-based treatment (FBT) for restrictive eating disorders. Clinicians who treat youth and accept Medicaid insurance within a predetermined group of participating California counties will be randomized to receive either online training or live two-day training in FBT. Data will be collected on the feasibility, acceptability, appropriateness, and effectiveness of the training (online vs. live). Following training, a subset of clinicians may opt into group consultation for one year. Consultation groups will be kept separate by training condition. Data will also be collected from clinicians on the extent to which they perceive the treatment itself (i.e., FBT) as feasible, acceptable, and appropriate for Medicaid-insured youth. In addition to implementation outcomes, de-identified clinical data will be collected from providers about their cases up to one year following the initial training.

ELIGIBILITY:
Inclusion Criteria:

* Mental health provider licensed to practice in the state of California, or unlicensed mental health providers in California who are formally employed by their agency/clinic and have a licensed clinical supervisor who agrees to take legal responsibility for any cases treated with FBT
* Must treat patients with Medicaid insurance in a participating county

Exclusion criteria:

- Students (practicum students, interns, externs) or other learners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin C Accurso, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: agency
Groups:
- Online Training: Online training will provide web-based training primarily focused on family-based treatment and appropriate adaptations to the treatment model. Interested participants who completed 100% of the online training were randomized to consultation groups (expert only vs. expert + peer consultation).
  Online training: Online training will be divided into training modules that will be completed by participants over the course of 6-8 weeks. Training will include didactic training videos, knowledge checks, example sessions, and a library of resources.
- Live Training: Live training will include two days of expert-led live training (via zoom). The content of the training will be similar to that provided in web-based training, primarily focused on family-based treatment and appropriate adaptations to the treatment model. Interested participants who completed 100% of the live training were randomized to consultation groups (expert only vs. expert + peer consultation).
  Live training: The live training will be delivered by two trainers over the course of two days via Zoom.
Period: Overall Study
Arm/Group | Online Training | Live Training
Started | 56; 16 agency | 29; 9 agency
Enrollment in Consultation | 33; 11 agency (Of the 33 online training participants who opted into consultation, 17 were assigned to expert consultation and 16 were assigned to expert + peer consultation.) | 10; 6 agency (Of the 10 online training participants who opted into consultation, all were assigned to expert consultation.)
Completed | 49; 16 agency | 21; 8 agency
Not Completed | 7; 0 agency | 8; 1 agency
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Online Training: Online training will provide web-based training primarily focused on family-based treatment and appropriate adaptations to the treatment model.
  Online training: Online training will be divided into training modules that will be completed by participants over the course of 6-8 weeks. Training will include didactic training videos, knowledge checks, example sessions, and a library of resources.
- Total: Total of all reporting groups
Arm/Group | Online Training | Live Training | Total
Number analyzed (Participants) | 56 | 29 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was available for 83 participants (online: n = 55, live: n = 28).
  years
    number analyzed (Participants) | 55 | 28 | 83
    (all) | 41.65 (9.26) | 37.39 (8.72) | 40.22 (9.25)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender female | 54 | 23 | 77
  Cisgender male | 2 | 4 | 6
  Gender non-binary or fluid | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 14 | 38
  Not Hispanic or Latino | 32 | 15 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 25 | 13 | 38
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 56 | 29 | 85
Primary discipline [Count of Participants; unit: Participants]
  Marriage/Family Therapy | 27 | 10 | 37
  Social Work | 20 | 15 | 35
  Psychology | 4 | 3 | 7
  Psychiatry | 2 | 0 | 2
  Other | 2 | 0 | 2
  Unknown | 1 | 1 | 2
Provide services in language other than English [Count of Participants; unit: Participants] | 33 | 15 | 48
Years clinical experience [Mean (Standard Deviation); unit: years] — Population: Clinical experience (years) was available for 82 participants (online: n = 54, live: n = 28).
  years
    number analyzed (Participants) | 54 | 28 | 82
    (all) | 9.78 (6.85) | 7.36 (5.68) | 8.95 (6.54)
Licensure status (licensed) [Count of Participants; unit: Participants] | 46 | 20 | 66
Any prior eating disorder treatment experience [Count of Participants; unit: Participants] | 29 | 14 | 43
Level of training and/or experience in FBT [Mean (Standard Deviation); unit: units on a scale] — Clinicians reported on the extent to which they had been exposed to or received training in FBT using a five-point scale (1 = no formal training or exposure, 2 = no formal training but some exposure, 3 = very little training, 4= moderate training, 5 = extensive training).
  units on a scale | 2.45 (1.21) | 2.03 (1.02) | 2.31 (1.16)
Training Preference [Count of Participants; unit: Participants]
  Online (strong preference) | 10 | 7 | 17
  Online (moderate preference) | 7 | 2 | 9
  Online (slight preference) | 4 | 2 | 6
  No preference | 8 | 6 | 14
  Live (slight preference) | 1 | 1 | 2
  Live (moderate preference) | 4 | 2 | 6
  Live (strong preference) | 22 | 9 | 31
Family-Based Treatment Knowledge Assessment (FBT-KA) [Mean (Standard Deviation); unit: score on a scale] — The Family-Based Treatment Knowledge Assessment (FBT-KA) is an 28-item measure that assesses knowledge about FBT for anorexia nervosa and atypical anorexia nervosa. The assessment focuses on general knowledge about FBT (e.g., contraindications, treatment phases), key principles (e.g., externalization, agnosticism, clinician as consultant), and key procedures (e.g., taking regular open weights). Scores range from 0 to 28, with higher scores indicating more knowledge.
  score on a scale | 8.30 (4.56) | 8.86 (4.57) | 8.49 (4.54)
Modified Practice Attitudes Scale (MPAS) [Mean (Standard Deviation); unit: score on a scale] — The Modified Practice Attitudes Scale (MPAS) is an eight-item measure with good reliability and validity that assesses clinician attitudes towards evidence-based treatments. Scores range from 0 to 32, with higher scores indicating more positive attitudes towards evidence-based practice. Population: MPAS data were available for 83 participants (online: n = 55, live: n = 28).
  score on a scale
    number analyzed (Participants) | 55 | 28 | 83
    (all) | 23.75 (3.48) | 22.21 (4.09) | 23.23 (3.74)
Organizational Readiness for Change (ORC-D4) [Mean (Standard Deviation); unit: score on a scale] — The Organizational Readiness for Change (ORC-D4) measure is a 30-item measure with acceptable reliability and validity that assesses attitudes, barriers, and facilitators within the working environment (e.g., collaboration and trust amongst peers, openness to change, management effectiveness). Scores range from 10 to 50, with higher scores indicating greater organizational capacity to implement a change. Population: ORC-D4 data were available for 82 participants (online: n = 54, live: n = 28).
  score on a scale
    number analyzed (Participants) | 53 | 27 | 80
    (all) | 36.23 (3.62) | 35.75 (3.46) | 36.06 (3.55)
Importance of eating disorders to organization [Mean (Standard Deviation); unit: units on a scale] — A five-item scale (extremely unimportant to extremely important) with a neutral mid-point was used to rank the extent to which eating disorders were perceived to be of importance to clinicians' organization (e.g., agency). Scores range from -2 to 2, with higher scores indicating greater importance. Population: Data on the importance of eating disorders in one's organization were available for 72 participants (online: n = 50, live: n = 22).
  units on a scale
    number analyzed (Participants) | 50 | 22 | 72
    (all) | 1.42 (0.93) | 1.23 (0.97) | 1.36 (0.94)
Importance of eating disorders to own practice [Mean (Standard Deviation); unit: units on a scale] — A five-item scale (extremely unimportant to extremely important) with a neutral mid-point was used to rank the extent to which eating disorders were important to clinicians' own practice. Scores range from -2 to 2, with higher scores indicating greater importance. Population: Data on the importance of eating disorders in one's own practice were available for 72 participants (online: n = 50, live: n = 22).
  units on a scale
    number analyzed (Participants) | 50 | 22 | 72
    (all) | 1.36 (0.90) | 1.23 (0.81) | 1.32 (0.87)
Comfort with eating disorders [Mean (Standard Deviation); unit: units on a scale] — A five-item scale (extremely uncomfortable to extremely comfortable) with a neutral mid-point was used to rank the degree to which clinicians feel comfortable treating EDs. Scores range from -2 to 2, with higher scores indicating greater comfort. Population: Data on comfort with eating disorders were available for 83 participants (online: n = 55, live: n = 28).
  units on a scale
    number analyzed (Participants) | 55 | 28 | 83
    (all) | -0.18 (1.16) | -0.25 (0.93) | -0.20 (1.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Training
Description: Training completion will be the number of participants who complete the full course of training.
Time Frame: Post-training (measured at the time of planned completion, which will be 10 weeks from the start of web-based training, or on the second day of live training)
Population: Data on training completion were available for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Online Training | Live Training
Number analyzed (Participants) | 56 | 29
Participants
  Completed training | 48 | 22
  Did not complete training | 8 | 7
Statistical Analysis 1: Comparison: Online Training vs Live Training; We used logistic multilevel models to examine the impact of training assignment (reference = live training) on training completion, with a random intercept at the agency level. Covariates included prior level of training and/or experience in FBT, attitudes towards evidence-based practice (MPAS), perceived importance of eating disorder treatment to organization, and training preference; Test type: Superiority; p = 0.47, Regression, Logistic; multilevel logistic regression; Odds Ratio (OR) = 0.617, 95% CI 2-sided [0.167 to 2.283]

2. Primary Outcome: Family-Based Treatment Knowledge Assessment (FBT-KA) Score at Post-Training
Description: The FBT Knowledge Assessment (FBT-KA) is an 28-item multiple-choice test that measures knowledge about FBT. Scores range from 0 to 28, with higher scores indicating more knowledge.
Time Frame: Baseline and post-training (measured immediately following completion of training)
Population: Data on post-training knowledge were available for 70 participants (online: n = 50, live: n = 20). However, all participants were included in the analysis. We used multiple imputation to account for missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Training | Live Training
Number analyzed (Participants) | 56 | 29
score on a scale | 20.52 (4.23) | 18.30 (2.96)
Statistical Analysis 1: Comparison: Online Training vs Live Training; We used linear multilevel models with restricted maximum likelihood (REML) estimation to examine the impact of training assignment (reference = live training) on knowledge acquisition at post-training, with a random intercept at the agency level. Covariates included baseline FBT-KA score, prior level of training and/or experience in FBT, attitudes towards evidence-based practice (MPAS), perceived importance of eating disorder treatment to organization, and training preference; Test type: Superiority; p = .29, Regression, Linear; multilevel linear regression with restricted maximum likelihood (REML) estimation; adjusted group difference unstandardized = -1.268, 95% CI 2-sided [-3.618 to 1.083]

3. Secondary Outcome: Number of Participants Who Receive FBT Consultation at 12 Months
Description: Providers will report on their receipt (yes/no) of FBT-specific consultation in the 12 months following completion of training.
Time Frame: 12-month follow-up (measured at 12 months from the deadline for completion of training)
Population: Data on 12-month engagement in consultation were available for 70 participants (online: n = 49, live: n = 21). However, all participants were included in the analysis. We used multiple imputation to account for missingness.
Measure: Count of Participants; unit: Participants
Arm/Group | Online Training | Live Training
Number analyzed (Participants) | 56 | 29
Participants
  Participating in FBT consultation | 28 | 10
  Not participating in FBT consultation | 21 | 11
  Unknown | 7 | 8
Statistical Analysis 1: Comparison: Online Training vs Live Training; We used logistic multilevel models to examine the impact of training assignment (reference = live training) on engagement in FBT consultation at 12 months, with a random intercept at the agency level. Covariates included baseline intent to seek FBT consultation, prior level of training and/or experience in FBT, attitudes towards evidence-based practice (MPAS), perceived importance of eating disorder treatment to organization, and training preference; Test type: Superiority; p = 0.92, Regression, Logistic; multilevel logistic regression; Odds Ratio (OR) = 1.160, 95% CI 2-sided [0.070 to 19.293]

ADVERSE EVENTS:
Time Frame: 15 months
Description: No serious adverse events were expected in this trial given that it was low-risk (i.e., providing behavioral health training to mental health clinicians).
Groups:
- Online Training: Online web-based training will provide online training primarily focused on family-based treatment and appropriate adaptations to the treatment model.
  Online training: Online web-based training will be divided into training modules that will be completed by participants over the course of 6-8 weeks. Training will include didactic training videos, knowledge checks, example sessions, and a library of resources.
Arm/Group | Online Training | Live Training
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/29
Other Adverse Events (participants affected / at risk) | 0/56 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT05389657/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05389657/ICF_001.pdf